CLINICAL TRIAL: NCT04218526
Title: Deep Brain Stimulation of the Cuneiform Nucleus for Levodopa-resistant Freezing of Gait in Parkinson's Disease
Acronym: DBS + FOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Jagid (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Jonathan Jagid, Associate Professor of Neurological Surgery, Neurology, Orthopedics, and Rehabilitation, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190702
Record Dates: First submitted 2019-12-02; First posted 2020-01-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Vercise DBS Group (Experimental): All participants will have the Vercise DBS system implanted.
  Interventions: Device: Vercise DBS System

INTERVENTIONS:
Device: Vercise DBS System — Vercise Deep Brain Stimulation (DBS) System that consists of two bilateral directional DBS Cartesia electrodes implanted in the cuneiform nucleus and a Gevia generator implanted in the upper chest area just below the clavicle.

SUMMARY:
The purpose of this research study is to determine if DBS is a safe and effective therapy for severe freezing of gait in patients with Parkinson's Disease. Freezing of gait (FOG) is a particularly debilitating motor deficit seen in a subset of patients with Parkinson's Disease (PD).

ELIGIBILITY:
Inclusion:

1. Confirmed Parkinson's Disease according to movement disorder neurologist with documented exclusion of other disorders such as fronto-temporal dementia (FTD)/ frontal gait disorder/normal pressure hydrocephalus (NPH)/progressive supranuclear palsy (PSP)
2. PD stage3 ON medication, with severe gait dysfunction and predominant axial symptoms: Movement Disorder Society-Unified Parkinson's Disease Rating Scale Tremor Dominant (MDS-UPDRS TD), Postural Instability Gait Difficulty (PIGD) ratio ≤ 0.90 and Freezing Of Gait Questionnaire (FOGQ) score > 12.
3. Age 40-75 with good response to Levodopa (defined as greater than 20% improvement in UPDRS score)
4. FOG refractory to LEVODOPA>600 mg
5. 6. Minimal tremor, bradykinesia, and rigidity symptoms, or well controlled with Levodopa and/or with already implanted STN/GPi DBS.
6. a) Poor candidate for STN or GPi DBS due to good control of tremor, bradykinesia, and rigidity symptoms with Levodopa b) or Post-operative STN/GPi DBS PD patients with significant residual non-levodopa responsive postural and gait instability
7. Must agree to full 6-month participation in study.

Exclusion:

1. Individuals with major executive dysfunction
2. Individuals with dementia, as defined by the Mattis Dementia Rating Scale-2 (DRS-2) score ≤ 130
3. Individuals with other neurocognitive impairments
4. Individuals who have depression, as defined for example by the Beck Depression Inventory II (BDI-II) > 25
5. Presence of major medical co-morbidities and other surgical contra-indications such as coagulopathy
6. Individuals who require diathermy, transcranial magnetic stimulation (TMS), or electroconvulsive therapy (ECT)
7. Individuals with a history of prior intracranial surgery
8. Individuals with a metallic implant in their head that is not MRI compatible (e.g., aneurysm clip, cochlear implant)
9. Individuals with active implantable devices anywhere in the body (e.g. cardiac pacemaker, defibrillator, spinal cord stimulator, implanted medication pump)
10. Individuals who are pregnancy or desire to become pregnant during the study
11. Individuals who are breastfeeding12.
12. Individuals who are on investigational drugs and any other intervention (not part of the guidelines for management of Parkinson's Disease) known to have a potential impact on outcome
13. Subjects utilizing recreational drugs at the time of screening will be excluded from the study with the exception of medicinal marijuana

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Percent Change in Gait Velocity | Baseline, 2 week, 6 weeks, 12 weeks, 24 weeks and 25-28 week post-op
  Percent change in gait velocity with and without bilateral cuneiform nucleus deep brain stimulation. Over a distance of 3 meters, gait velocity will be measured using the timed Up and Go test instrumented with Mobility Lab accelerometers.
Percent change in UPDRS Part III on/off stimulation | Baseline, 2 week, 6 weeks, 12 weeks, 24 weeks and 25-28 week post-op
  Percent change in Unified Parkinson's Disease Rating Scale (UPDRS) Part III on/off stimulation across study visits relative to pre-operative assessment

SECONDARY OUTCOMES:
Percent Change in FOG Questionnaire | Baseline, 2 week, 6 weeks, 12 weeks, 24 weeks and 25-28 week post-op
  Freezing of Gait (FOG) Questionnaire is a 6-item questionnaire with each item scored from 0-4. The total score ranges from 0-24 with the higher score indicating more severe freezing of gait .
Percent Change in PDQ 39 | Baseline, 2 week, 6 weeks, 12 weeks, 24 weeks and 25-28 week post-op
  Parkinson's Disease Questionnaire (PDQ-39) is 39-item questionnaire with a total score ranging from 0-156 with the higher score indicating poorer quality of life.
Percent Change in PDQ-L | Baseline, 2 week, 6 weeks, 12 weeks, 24 weeks and 25-28 week post-op
  Parkinson's Disease Quality of Life Questionnaire is a 37-item questionnaire with a total score ranging from 0-185 with the higher score indicating poorer quality of life.
Percent Change in Muscle Amplitude | Baseline, 24 weeks
  Percent change in muscle amplitude during gait testing using electromyography (EMG)
Percent Change in number of Falls | Baseline, 24 weeks
  Percent change in number of falls during gait testing sessions and on item 13 of UPDRS III (falls unrelated to freezing)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan R Jagid, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang SJ, Cajigas I, Guest JD, Noga BR, Widerstrom-Noga E, Haq I, Fisher L, Luca CC, Jagid JR. MR Tractography-Based Targeting and Physiological Identification of the Cuneiform Nucleus for Directional DBS in a Parkinson's Disease Patient With Levodopa-Resistant Freezing of Gait. Front Hum Neurosci. 2021 Jun 8;15:676755. doi: 10.3389/fnhum.2021.676755. eCollection 2021. PMID 34168545
- [Derived] Chang SJ, Cajigas I, Guest JD, Noga BR, Widerstrom-Noga E, Haq I, Fisher L, Luca CC, Jagid JR. Deep brain stimulation of the Cuneiform nucleus for levodopa-resistant freezing of gait in Parkinson's disease: study protocol for a prospective, pilot trial. Pilot Feasibility Stud. 2021 Jun 2;7(1):117. doi: 10.1186/s40814-021-00855-7. PMID 34078477